CLINICAL TRIAL: NCT06403748
Title: Evaluation of the Effect of a Food Supplementation With a Combined Food Supplement on Lipid Pattern, Indexes of NAFLD and Systemic Inflammation in Healthy Subjects With Suboptimal LDL-C Levels: a Two-arm Double-blind, Placebo-controlled, Randomized, Clinical Trial
Brief Title: Effect of a Dietary Supplement on Lipid Pattern, Indexes of NAFLD and Systemic Inflammation in Healthy Subjects With Suboptimal LDL-C Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Prof. Dr., University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NUT1-BO-2022
Record Dates: First submitted 2024-03-09; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hypercholesterolemia; Inflammation
MeSH Terms: conditions — Hypercholesterolemia; Inflammation | interventions — dan-shen root extract; Folic Acid; Chromium; Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement (Active Comparator)
  Interventions: Dietary Supplement: Dietary supplement formulated with components of natural origin: artichoke, danshen, bergamot, folic acid, chromium and excipients.
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary supplement formulated with components of natural origin: artichoke, danshen, bergamot, folic acid, chromium and excipients. — The study will be conducted in male and female subjects, at least 18 and less than 70 years of age, with suboptimal level of LDL-Cholesterol (LDL 115-190 mg/dL) randomized into two groups to receive a preconstituted food supplement (NUT) combination containing (Red yeast rice 160 mg + Berberis aristate 449,7 mg + Folic acid 200 μg and others) in combination with a standard Mediterranean diet at low cholesterol content (<200 mg/day) (Standard of Care - SOC) [group 1], or a PLACEBO in combination with hypo-cholesterol diet (healthy Mediterranean diet following the indication of the European Atherosclerosis Society guidelines) [group 2].
  Arms: Dietary supplement
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of our research will be to evaluate if, in subjects with a low-moderate cardiovascular risk (CV risk>1% but < 5%) evidenced by sub-optimal cholesterol levels as per ESC/EAS guidelines (LDL cholesterol >115 mg/dL, < 190 mg/dL) supplementation with a food supplement is able to significantly influence plasma lipid levels. Furthermore, the systemic activation status of the inflammatory cascade and the arterial wall stiffness will be investigated.

ELIGIBILITY:
Inclusion Criteria:

The subjects will have to meet all the following inclusion criteria:

1. Subjects agree to participate in the study and having dated and signed the informed consent form.
2. Male or female aged ≥ 18 years and ≤ 70 years old.
3. LDL-Cholesterol plasma levels >115 mg/dL and < 190 mg/dL.
4. TG<400 mg/dL.
5. Subjects who, according to the SCORE charts, have a low or moderate cardiovascular risk (defined as a total cardiovascular risk < 5%) and for whom, according to ESC/EAS guidelines 2012, the intervention strategy does not require a pharmacological lipid- lowering intervention.
6. Subjects who have the capability to communicate, to make themselves understood, and to comply with the study's requirements.

Exclusion Criteria:

Subjects fulfilling one or more of the following exclusion criteria will not be included in the study:

1. Subjects already affected by cardiovascular diseases (secondary prevention) or with estimated 10 years cardiovascular disease risk > 5%;
2. Obesity (BMI>30 kg/m2) or diabetes mellitus;
3. Assumption of lipid-lowering drugs or food supplements, or drugs potentially affecting the lipid metabolism;
4. Antihypertensive treatment not stabilized for at least 3 months;
5. Anticoagulant therapy
6. Uncontrolled hypertension (systolic blood pressure> 190 mmHg or diastolic arterial pressure> 100 mmHg);
7. Known current thyroid, gastrointestinal or hepatobiliary diseases;
8. Any medical or surgical condition that would limit the participant adhesion to the study protocol;
9. Abuse of alcohol or drugs (current or previous);
10. History of malignant neoplasia in the 5 years prior to enrolment in the study;
11. History or clinical evidence of inflammatory diseases such as severe arthritis, systemic lupus erythematosus or chronic inflammatory diseases or current therapy with immunosuppressive agents or long-term glucocorticoids;
12. History or clinical evidence of any significant concomitant disease that could compromise the safety of the subject or the possibility of completing the study;
13. Known previous intolerance to one component of the tested nutraceuticals or to one of these plant species: Asteraceae or Compositae;
14. Women in fertile age not using consolidated contraceptive methods
15. Pregnancy and Breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2024-10-11 (Estimated); Study Completion 2024-10-11 (Estimated)

PRIMARY OUTCOMES:
Effect of the dietary supplement on LDL-C at 6-week follow-up | 6 weeks
  The primary objective is to compare the effect on LDL-C after 6 weeks of treatment with a combined food supplement compared to placebo (standard diet only).
Effect of the dietary supplement on LDL-C at 6-week follow-up | 12 weeks
  The primary objective is to compare the effect on LDL-C after 12 weeks of treatment with a combined food supplement compared to placebo (standard diet only).

SECONDARY OUTCOMES:
Effect of the dietary supplement on lipid fractions | 12 weeks
  Evaluate the effect of the tested combined food supplement intake on changes in other lipid fractions
Effect of the dietary supplement on apolipoproteins | 12 weeks
  Evaluate the effect of the tested combined food supplement intake on changes in apolipoproteins
Effect of the dietary supplement on hsCRP | 12 weeks
  Evaluate the effect of the tested combined food supplement intake on hsCRP levels
Effect of the dietary supplement on indexes of NAFLD | 12 weeks
  Evaluate the effect of the tested combined food supplement intake on validated indexes of non-alcoholic fatty liver disease
Effect of the dietary supplement on waist circumference | 12 weeks
  Evaluate the effect of the tested food supplement intake on changes in waist circumference. Waist circumference will be measured in a horizontal plane at the end of a normal expiration, at the midpoint between the inferior margin of the last rib and the superior iliac crest.
Effect of the dietary supplement on weight | 12 weeks
  Evaluate the effect of the tested food supplement intake on changes in weight. Weight will be measured to the nearest 0.1 Kg.
Effect of the dietary supplement on blood pressure | 12 weeks
  Evaluate the effect of the tested food supplement intake on changes in systolic blood pressure and diastolic blood pressure
Effect of the dietary supplement on creatininemia | 12 weeks
  Evaluate the effect of the tested food supplement intake on changes in creatininemia
Effect of the dietary supplement on eGFR | 12 weeks
  Evaluate the effect of the tested food supplement intake on renal function, evaluated as eGFR
Effect of the dietary supplement on CPK levels | 12 weeks
  Evaluate the effect of the tested food supplement intake on changes in the blood levels of CPK
Tolerability of the dietary supplement | 12 weeks
  Comparative evaluation of the short-term tolerability of the tested food supplement. Tolerability will be evaluated through a continuous monitoring during the study, to detect any adverse event, clinical safety, laboratory findings, vital sign measurements, and physical examinations
Acceptability of the dietary supplement | 12 weeks
  Comparative evaluation of the short-term acceptability of the tested food. Acceptability will be evaluated by the use of a 10-point hedonic scale, where 1 = Disliked extremely and 9 = Liked extremely.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No